CLINICAL TRIAL: NCT06268756
Title: Fear of Other's Judgment, Self-esteem and Use of Social Networks Among Students
Acronym: RESANXIEST
Status: Recruiting | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_020_RESANXIEST
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Self-esteem
Keywords: Fear of judgment; self-esteem; social networks; student
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: students
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Fear of being judged negatively by others can lead to avoidance of social situations or even social isolation. If the intensity of this fear is excessive and results in significant impairment of functioning or significant suffering, the subject may suffer from social anxiety.

The considerable growth of social networks in a decade has led to the emergence of new behaviors among young people. Individuals spend on average 2 hours and 27 minutes per day with differences in usage: time spent, social network used, function sought. The use of these networks may be reasonable and moderate but may also be excessive and abusive (Amnon, 2014). Some authors even talk about addiction or dependence on social networks (Perales and Billieux, 2020) even if the existence of this disorder is not consensus.

People who fear being judged negatively by others may be more at risk of misuse of social networks. Indeed, the use of social networks would compensate for their existing problems (Kardefelt-Winther, 2014) and would thus be a new emotional management strategy. It would also reduce dreaded social situations such as face-to-face exchanges (Weidman and Rodebaugh, 2012; Yen and Ko, 2012). Self-esteem is defined as a subjective judgment of oneself in relation to one's values and vision of the real and ideal self (Rosenberg. 1979). The greater the gap between the vision of the real self and the ideal self, the lower the self-esteem.

DETAILED DESCRIPTION:
The objective of the study is to study the influence of self-esteem on the association between the fear of being judged negatively by others and the use of social networks.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* students at a French school or university
* using social media
* agreeing to participate in the study

Exclusion Criteria:

* Protected by law
* Refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: students using social networks
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-04-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self-esteem Scale | Day 0
  a self-administered questionnaire containing ten statements measuring a person's general attitude towards his own worth. For each, the subject indicates his or her agreement on a Likert scale from 1 to 4, with 1 meaning "strongly disagree", 2 "somewhat disagree", 3 "somewhat agree" and 4 "strongly agree".
  The score is interpreted as follows:
  * A score below 25 indicates very low self-esteem.
  * A score between 25 and 31 indicates low self-esteem.
  * A score between 31 and 34 indicates average self-esteem.
  * A score between 34 and 39 indicates high self-esteem.
  * A score above 39 indicates very high self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: JULIEN SWEERTS Sabrina, Study Director — Université de Reims Champagne-Ardenne
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided